CLINICAL TRIAL: NCT04001530
Title: Verification of Half Normal Saline as a Superior Irrigant in the Catheter Radiofrequency Ablation of Typical Cavotricuspid Isthmus Dependent Atrial Flutter: A Multicenter Study
Brief Title: Half-normal Saline in Atrial Flutter Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Benedict Glover, Staff electrophysiologist Schulich Heart Program, Associate Professor University of Toronto, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 156-2019
Record Dates: First submitted 2019-06-26; First posted 2019-06-28 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-07

CONDITIONS: Atrial Flutter
MeSH Terms: conditions — Atrial Flutter | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Half-normal saline (Experimental): Use of half-normal saline (0.45% NaCl) as an irrigant for open-irrigated ablation catheters
  Interventions: Drug: Half Normal Saline 0.45% Infusion Solution Bag
- Normal saline (Active Comparator): Use of normal saline (0.9% NaCl) as an irrigant for open-irrigated ablation catheters
  Interventions: Drug: Normal Saline 0.9% Infusion Solution Bag

INTERVENTIONS:
Drug: Half Normal Saline 0.45% Infusion Solution Bag — Randomization to half normal saline
  Arms: Half-normal saline
Drug: Normal Saline 0.9% Infusion Solution Bag — Randomization to normal saline
  Arms: Normal saline

SUMMARY:
To assess the acute and long-term efficacy of half-normal saline compared to normal saline for irrigation of open-irrigated catheters during catheter ablation for the treatment of cavotricuspid isthmus dependent atrial flutter.

DETAILED DESCRIPTION:
It is unclear whether ionic strength affects energy delivery and ablation lesion size during radiofrequency ablation for atrial flutter. Given that saline contains ionic sodium and chloride in the solution, it has conductive properties that may disperse radiofrequency energy away from the tip-tissue interface, thereby reducing current density and lesion size compared to ablation with nonionic solutions. The efficacy of half-normal saline will be measured by the time taken to create bidirectional block across the cavotricuspid isthmus as well as the acute recurrence rate within 30 minutes of the initial occurrence of bidirectional block and the 1 year freedom from flutter recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age at the time of enrollment
* Patients presenting for right sided typical atrial flutter ablation who have a clinical indication to undergo catheter ablation
* Fully informed written informed consent by either the subject or subject's legal representative and ability for subject to comply with study responsibilities

Exclusion Criteria:

* The presence of thrombus within the left atrial appendage
* Prior catheter ablation of the cavotricuspid isthmus for right sided atrial flutter
* The inability to provide consent or comply with study requirements
* A predicted life expectancy of < 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Time taken to produce bidirectional block | intraprocedural
Acute recurrence rate < 30 minutes of initial occurrence of bidirectional block | intraprocedural
Freedom from atrial flutter recurrence | 1 year

SECONDARY OUTCOMES:
Time taken for termination of atrial flutter | intraprocedural
Total radiofrequency ablation time and procedural time | intraprocedural

OTHER OUTCOMES:
Incidence of procedure-related complications | at the time of the procedure and up to 1 month
  pericardial effusion due to cardiac perforation or pericarditis, transient ischemic attack/stroke, systemic embolism, phrenic nerve injury, pulmonary vein stenosis, atrio-esophageal fistula, death
Incidence of steam pops | periprocedural
  marker of excessive heating of the tissue

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Multicentre study, patient data deidentified for post-enrolment analysis